CLINICAL TRIAL: NCT04178785
Title: Remifentanil Versus Fentanyl During Laparoscopic Hysterectomy- a Randomized Control Trial
Brief Title: Remifentanil Versus Fentanyl During Laparoscopic Hysterectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0038-19-WOMC
Record Dates: First submitted 2019-10-22; First posted 2019-11-26 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Anesthesia
Keywords: laparoscopic; remifentanil; fentanyl; hysterectomy
MeSH Terms: interventions — Remifentanil

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- REMIFENATIL (Active Comparator): Prospective, single-center single blind randomized controlled trial. Patients electively admitted for laparoscopic hysterectomy will be approached for requirement. After obtaining a written informed consent, patients will be randomly assigned either to the study group (Remifentanil group) or to the control group (Fentanyl group) in a 1:1 ratio. A blocked randomization scheme will be created using a computer-generated list of random numbers.
  Interventions: Drug: Remifentanil
- FENTANYL (No Intervention): Prospective, single-center single blind randomized controlled trial. Patients electively admitted for laparoscopic hysterectomy will be approached for requirement. After obtaining a written informed consent, patients will be randomly assigned either to the study group (Remifentanil group) or to the control group (Fentanyl group) in a 1:1 ratio. A blocked randomization scheme will be created using a computer-generated list of random numbers.

INTERVENTIONS:
Drug: Remifentanil — Patients electively admitted for laparoscopic hysterectomy will be approached for requirement. After obtaining a written informed consent, patients will be randomly assigned either to the study group (Remifentanil group) or to the control group (Fentanyl group) in a 1:1 ratio.
  Arms: REMIFENATIL

SUMMARY:
Introduction- During laparoscopic procedures surgical field exposure is one of the crucial aspects for a successful surgery. Exposure can be optimized by pneumoperitoneum, positioning of the patient and muscle relaxation.

The European Association for Endoscopic Surgery has recommended using the lowest intraperitoneal pressure allowing adequate exposure of the operative field rather than using a routine pressure. A way to lower intraabdominal pressure during laparoscopic procedures is to employ a deeper level of neuromuscular blockade.

Intravenous (IV) opioids such as fentanyl and remifentanil are commonly used to provide analgesia and supplement sedation during general anesthesia.

In terms of analgesia, management of intraoperative stress, remifentanil exhibits similar effects to fentanyl in adult healthy volunteers and surgical patients.

In clinical practice, if the surgeon asks for relaxation toward the end of the surgery, then many anesthesiologists will increase the dose of the IV opioids. In our experience the use of remifentanil achieves a better muscle relaxation and surgical space exposure with a lower intraabdominal pressure and less need for a neuromuscular blockage as compared to fentanyl.

Thus, the investigators aimed to compare the use of fentanyl versus remifentanil during laparoscopic hysterectomy. Because surgical complications due to inadequate exposure are a rare event, the typical way to study this issue is to use surgeon's satisfaction score.

DETAILED DESCRIPTION:
Study design- Prospective, single-center single blind randomized controlled trial. Patients electively admitted for laparoscopic hysterectomy will be approached for requirement. After obtaining a written informed consent, patients will be randomly assigned either to the study group (Remifentanil group) or to the control group (Fentanyl group) in a 1:1 ratio. A blocked randomization scheme will be created using a computer-generated list of random numbers.

study protocol-

1. anesthesia is induced and maintained with propofol
2. Ventilation is performed with volume/pressure control mode with a tidal volume of 6-8 ml/kg, a frequency of 10-12/min and a positive end-expiratory pressure of 5 cm H2O aiming at normocapnia.
3. Tracheal intubation is performed 2 min after administration of the muscle relaxant 0.6-1.2 mg/kg rocuronium.
4. Patients in the study group will receive 0.2 mcg/kg/min Remifentanil
5. Fentanyl at the dose of 100mcg will be administered to all the patients in the control group
6. The gynecologist, surgical staff and patients will be blinded to group allocation.
7. During surgery additional muscle relaxant will be given only when asked by the gynecologist and will be mentioned in the anesthesiologic chart
8. The investigator managed the insufflation of the abdomen to 12 mmHg pneumoperitoneum.
9. Patients will be placed in the lithotomy position in a 30-degree head-down body position.
10. Antibiotic prophylaxis is given for all patients
11. The gynecologists will evaluate the surgical conditions before a colpotomy is made in a circumferential fashion around the cervix and toward the end of the surgery on four-point rating scale (1: excellent, 2: good, 3: acceptable 4: poor)
12. The gynecologists will also rate surgical space conditions on a numeric rating scale (NRS), where NRS 0 indicated optimal surgical space conditions and NRS 100 indicated unacceptable surgical space conditions and an intervention is needed to secure acceptable surgical space6

ELIGIBILITY:
Inclusion Criteria:

* age >18
* scheduled for laparoscopic hysterectomy

Exclusion Criteria:

* known allergy to medications that are included in the trial, severe renal disease or impaired liver function

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 76 (Estimated)
Dates: Start 2019-10-22 (Actual); Primary Completion 2020-10-22 (Estimated); Study Completion 2020-11-01 (Estimated)

PRIMARY OUTCOMES:
Surgical space conditions with modification of a 4-point scale. AT TIME OF COLPOTOMY | through study completion, an average of 1 year
  1. grade 1 (optimal) = optimal surgical space conditions;
  2. grade 2 (good) = nonoptimal conditions, but an intervention was not considered;
  3. grade 3 (acceptable) = an intervention was considered to improve surgical space;
  4. grade 4 (poor) = inadequate conditions and an intervention was necessary to ensure acceptable surgical space.
Surgical space conditions with modification of a 4-point scale. AT THE END OF SURGERY | through study completion, an average of 1 year
  1. grade 1 (optimal) = optimal surgical space conditions;

SECONDARY OUTCOMES:
surgical space conditions on a numeric rating scale (NRS) | through study completion, an average of 1 year
  where NRS 0 indicated optimal surgical space conditions and NRS 100 indicated unacceptable surgical space conditions and an intervention is needed to secure acceptable surgical space

CONTACTS AND LOCATIONS:
Locations (1):
- Wolfson medical center, Holon, Israel